CLINICAL TRIAL: NCT06305611
Title: Comparison and Performance of Kobayashi and Kawanet IVIg Resistance Scores in a Multi-centric European and North Indian Cohort of KaWasaki dIsease (the KIWI Study)
Brief Title: European and North Indian Cohort of KaWasaki dIsease
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Gabriele Simonini, MD, Meyer Children's Hospital IRCCS
Other Study IDs: KIWI
Record Dates: First submitted 2024-02-16; First posted 2024-03-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kawasaki disease (KD) is currently the leading cause of acquired heart diseases in children in developed countries. Cardiac involvement is the main determinant of the long-term prognosis of these patients, as coronary aneurisms (CAAs) may lead to ischemic heart disease and even sudden death. The current standard of care for KD has consistently reduced CAAs frequency from 25-30% to about 5%. Unfortunately, 10-20% of KD patients results resistant to standard treatment leading to a major risk of cardiac complications. Thus, scoring systems have been constructed in order to identify patients likely to be resistant to IVIG and who may benefit from more aggressive initial therapy. Different scoring scales developed by Kobayashi, Egami et Sano had shown a good sensitivity (77-86%) and specificity (67-86%) in predicting IVIG unresponsiveness in Japanese populations. However, their predictive value was not confirmed by subsequent studies in different ethnic populations. Recently, the French Kawanet group have proposed a IVIG unresponsiveness score that provided good sensitivity and acceptable specificity in a non-Asian KD population even if it was not subsequent validated by an external study. In our study population, the achievement of specificity and sensitivity values for both scores consistent with those reported by the original studies (sensitivity 70% and specificity 80% for Kobayashi and sensitivity 77% and specificity 60% for Kawanet), will be considered a success.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than 18 years at diagnosis
* Diagnosis of KD according to the AHA criteria

Exclusion Criteria:

* Patients who do not meet the criteria for KD
* Patients for which an alternative infectious diagnosis was not investigated and/or excluded.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The setting is represented by 1 Asian and 4 European pediatric rheumatology centres which with internationally recognized expertise in the treatment and follow-up of a large number of Kawasaki disease patients
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
IVIG resistance rate | through study completion, an average of 1 year
  IVIG resistance rate in patients with KD and stratification according to different ethnic groups.
percentage of IVIG-resistant patients | through study completion, an average of 1 year
  percentage of IVIG-resistant patients who met the Kobayashi and KAWANET criteria, and specificity and sensitivity of the criteria within the different ethnic groups.

CONTACTS AND LOCATIONS:
Locations (27):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil
- Croatia (2):
  - Children's Hospital Zagreb, Zagreb
  - University Hospital Centre Zagreb, University School of Medicine, Zagreb
- Le Kremlin-Bicetre University Hospital, Paris-Sud University - CEREMAI, Le Kremlin-Bicêtre, France
- India (6):
  - Manipal Hospital, Bangalore
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Sri Ramachandra Medical Centre, Chennai
  - Amrita Institute of Medical Sciences, Kochi
  - Institute of Child Health, Kolkata
  - Vivekananda Institute of Medical Sciences, Kolkata
- Meir Medical Centre, Kfar Saba, Israel
- Italy (8):
  - ASST Papa Giovanni XXIII, Bergamo
  - Spedali Civili, Brescia
  - Meyer Children's Hospital IRCCS, Florence
  - IRCCS Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico, Milan
  - P.O. "Giovanni Di Cristina", Palermo
  - Università di Torino, Torino
  - IRCCS Burlo Garofolo, Trieste
- Beatrix Kinderkliniek, University Medical Center, Groningen, Netherlands
- Spain (2):
  - Hospital de Sabadell, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
- Chiang Mai University Hospital, Chiang Mai, Thailand
- Turkey (Türkiye) (3):
  - Hacettepe University Children's Hospital, Ankara
  - Health Sciences University, Umraniye Education and Research Hospital, Istanbul
  - Istanbul Uni. Istanbul Med.Fac, Istanbul
- Royal Hospital for Children, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No